CLINICAL TRIAL: NCT07094815
Title: Comparative Outcomes of Uterus-Preserving and Hysterectomy Approaches in Laparoscopic Lateral Suspension
Brief Title: Effectiveness of Laparoscopic Lateral Suspension With or Without Hysterectomy in Pelvic Organ Prolapse
Acronym: LLS-HYS
Status: Completed | Type: Observational
Sponsor: Havva Betül Bacak (Other Government)
Responsible Party: Sponsor-Investigator, Havva Betül Bacak, M.D, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Other Study IDs: lateralsuspwithuterusornot
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Organ Prolapse (POP); Uterine Prolapse
Keywords: Laparoscopic Lateral Suspension; Uterus Preservation; Uterine Prolapse; Pelvic Organ Prolapse; Minimally Invasive Surgery; POP-Q System; Surgical Outcomes; Gynecologic Surgery; Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LLS with Hysterectomy: Patients who underwent laparoscopic lateral suspension combined with total laparoscopic hysterectomy.
- Uterus-Preserving LLS: Patients who underwent laparoscopic lateral suspension with uterine preservation.

SUMMARY:
This study aims to compare the effectiveness of laparoscopic lateral suspension (LLS) with and without hysterectomy in the treatment of pelvic organ prolapse. Pelvic organ prolapse is a condition that affects many women and can significantly reduce quality of life. Laparoscopic lateral suspension is a minimally invasive surgical technique used to correct this condition. In some cases, the uterus is preserved, while in others, hysterectomy is performed at the same time.

The study retrospectively evaluates patients who underwent laparoscopic lateral suspension, either with or without hysterectomy, at SBÜ Gaziosmanpaşa Training and Research Hospital. Medical records were reviewed to collect information about surgery duration, anatomical success (measured by the POP-Q system), complication rates, blood loss, hospital stay, and recurrence rates.

The goal of this study is to determine whether performing a hysterectomy during laparoscopic lateral suspension has a significant effect on surgical outcomes. The findings may help guide surgical decision-making and improve treatment strategies for women with pelvic organ prolapse.

DETAILED DESCRIPTION:
This retrospective cohort study was conducted at SBÜ Gaziosmanpaşa Training and Research Hospital to compare the outcomes of laparoscopic lateral suspension (LLS) with and without concomitant hysterectomy in women with pelvic organ prolapse (POP). POP is a prevalent condition that significantly affects quality of life, and LLS is increasingly performed as a minimally invasive approach that allows either uterine preservation or hysterectomy.

A total of 87 patients treated between 2021 and 2024 were analyzed: 43 underwent LLS with total laparoscopic hysterectomy, and 44 underwent uterus-preserving LLS. Preoperative, intraoperative, and postoperative data were collected from electronic medical records, operative reports, and follow-up documentation, with at least 12 months of follow-up. Outcome measures included POP-Q scores, operative time, blood loss, hospital stay, perioperative complications, recurrence, pelvic pain, and urinary incontinence.

The analysis showed that both groups achieved significant anatomical improvement, with no significant differences in recurrence, pelvic pain, or urinary incontinence. However, hysterectomy was associated with longer operative times, increased blood loss, and longer hospital stays. Vaginal length was better preserved in uterus-preserving procedures. No major intraoperative or postoperative complications occurred.

These findings indicate that adding hysterectomy to LLS increases surgical burden without conferring additional anatomical or functional benefit. Uterus-preserving LLS appears to be a safe and effective option in appropriately selected patients, supporting shared decision-making in pelvic reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 40 to 80 years
* Diagnosis of pelvic organ prolapse (POP) requiring surgical management
* Underwent laparoscopic lateral suspension (LLS) with or without concomitant total laparoscopic hysterectomy
* Minimum of 12 months postoperative follow-up available
* Ability to provide informed consent for use of medical data in this retrospective study

Exclusion Criteria:

* History of connective tissue disorders
* History of prior pelvic reconstructive surgery
* Active pelvic infection or suspected malignancy at the time of surgery
* Severe systemic disease that could significantly affect surgical outcomes
* Incomplete medical records or missing follow-up data

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 40 to 80 years who underwent laparoscopic lateral suspension (LLS) with or without concomitant total laparoscopic hysterectomy for the treatment of pelvic organ prolapse at SBÜ Gaziosmanpaşa Training and Research Hospital between 2021 and 2024. All patients had at least 12 months of postoperative follow-up, and data were collected retrospectively from medical records.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Anatomical Success Based on POP-Q System | 12 months after surgery
  Primary Outcome Title:
  Number of Participants Achieving Anatomical Success Based on POP-Q System
  Description:
  Anatomical success is defined as all assessed POP-Q points (Aa, Ba, C, D, Ap, Bp) being at or above -1 cm (no prolapse extending more than 1 cm below the hymen).
  POP-Q scale values: Negative values indicate the point is above the hymen (better anatomy), positive values indicate prolapse below the hymen (worse anatomy).
  Typical range: Aa, Ba, Ap, Bp = -3 to +3 cm; C and D vary according to total vaginal length (TVL).
  Time Frame:
  12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Gaziosmanpaşa Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study is based on retrospective medical record review and no consent for data sharing was obtained from participants. All data are stored and analyzed internally according to institutional policies and ethical approvals.

REFERENCES:
- [Background] Kumbasar S, Salman S, Sogut O, K Gencer F, Bacak HB, Tezcan AD, Timur GY. Uterine-sparing laparoscopic lateral suspension in the treatment of pelvic organ prolapse. J Obstet Gynaecol Res. 2023 Jan;49(1):341-349. doi: 10.1111/jog.15459. Epub 2022 Oct 5. PMID 36196844